CLINICAL TRIAL: NCT02832297
Title: Prospective Outcomes Study: Vectra® DA Guided Care Compared to Usual Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Crescendo Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 088-CL-01
Record Dates: First submitted 2016-07-07; First posted 2016-07-14 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2017-07

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vectra DA (Arm A) (Other): Treatment intensification with non-biologic DMARDS guided by Vectra DA
  Interventions: Other: Vectra DA
- Usual care (Arm B) (Other): Treatment intensification by usual care without using Vectra DA
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Vectra DA
  Arms: Vectra DA (Arm A)
Other: Usual Care
  Arms: Usual care (Arm B)

SUMMARY:
In this 12-month multi-center prospective, site-randomized, two-arm trial, approximately 318 biologic-naïve subjects with RA who are candidates for treatment intensification due to inadequate response to MTX monotherapy will be enrolled at up to 60 study sites.

DETAILED DESCRIPTION:
To determine whether a strategy of Vectra DA guided care (Arm A), compared with usual care (Arm B), achieves non-inferior clinical outcomes while reducing the cost of treatment in patients with active RA and an inadequate response to MTX monotherapy.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible to participate in the study if they meet all the following criteria:

1. Willing and able to sign an ICF
2. Age 18 to 80 years at enrollment
3. Meets the 2010 ACR/EULAR criteria and/or 1987 criteria for RA, as determined by a board-certified rheumatologist ≥3 months prior to enrollment
4. Received uninterrupted treatment with weekly MTX begun ≥3 months prior to enrollment, at a stable dose of ≥15 mg per week for at least 4 weeks prior to enrollment. A history of therapy with split dose oral MTX or parenteral MTX is acceptable only if the weekly MTX dose was always ≤20 mg/week during the 3 months prior to enrollment.
5. CDAI >10 as assessed by the Investigator at screening
6. At least 3 swollen joints (SJC ≥3) and 3 tender joints (TJC ≥3) out of 28 joints as assessed by the Investigator at screening
7. Must be eligible for treatment intensification with non-biologic and biologic DMARDs
8. Documented evidence of seropositivity (RF and/or anti-CCP antibodies). Seronegative subjects are allowed if erosive disease attributable to RA is documented on X-rays.

Exclusion Criteria:

Subjects will be ineligible to participate in the study if they meet any of the following criteria:

1. Use of a non-biologic DMARD other than MTX within 3 months prior to enrollment
2. MTX administered SQ or as an oral split dose at >20 mg/week any time during the 3 months prior to enrollment
3. Two or more DMARDs used in combination (i.e., concomitantly), including but not limited to: MTX, HCQ, SSZ, LEF, cyclosporine, azathioprine, gold or penicillamine any time prior to enrollment
4. Biologic DMARD or JAKi use any time prior to enrollment
5. Any contraindication to use of MTX, HCQ, LEF or biologic DMARDs
6. Opiate use during the 2 weeks prior to enrollment
7. Oral corticosteroids during the month prior to enrollment at a dosage >10 mg/day prednisone (or equivalent) or at a non-stable dose ≤10 mg/day prednisone (or equivalent)
8. MTX intolerance prior to enrollment that limits its use
9. Inflammatory joint disease (other than RA) or any other systemic autoimmune disorder. (Osteoarthritis is not a basis for exclusion.)
10. Primary or secondary immunodeficiency
11. Active infection (excluding fungal infection of nail beds); or acute or chronic infection requiring hospitalization or treatment with parenteral systemic antibiotics within one month of enrollment or treatment with oral antibiotics within 2 weeks of enrollment
12. IA, intravenous or IM corticosteroids during the month prior to enrollment
13. Initiation or non-stable dosing of NSAIDs within 2 weeks prior to enrollment
14. Vectra DA testing within 3 months prior to enrollment
15. Live vaccine within 90 days of enrollment
16. Active substance abuse or psychiatric illness likely to interfere with protocol conduct
17. History of severe allergic or anaphylactic reaction to any monoclonal antibody therapy
18. Known infection with HIV (HIV testing will not be a requirement for trial entry); a past or current history of hepatitis B virus or hepatitis C virus infection
19. History of malignancy within the past five years or any evidence of persistent malignancy, except fully excised basal cell or squamous cell carcinomas of the skin, or cervical carcinoma in situ that has been treated or excised in a curative procedure
20. Pregnancy or inadequate contraception in women of childbearing potential
21. Breast feeding or lactating
22. Medical, psychiatric, cognitive or other conditions that, in the opinion of the Investigator, may compromise the ability of the subject to understand the study information, to give informed consent, to comply with the trial protocol, or to complete the study
23. Presently enrolled in another clinical trial
24. Vectra DA score at screening that is outside the applicable range as required for subject enrollment

Note: Screening for TB is not required for subjects participating in the study. If an Investigator is considering a subject for treatment with a biologic DMARD in the study, guidelines for TB screening need to be followed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change in DAS28 at Month 6 | Baseline to 6 months
Percentage of subjects using any biologic DMARD or JAK inhibitor to Month 6 | Baseline to 6 months

SECONDARY OUTCOMES:
Percentage of subjects with ACR20 response at Month 6 | Baseline to 6 months
Change in HAQ-DI score at Month 6 | Baseline to 6 months
Percentage of subjects with radiographic non-progression at 12 months | Baseline to 12 months
  Radiographic non-progression will be defined as change in modified total Sharp score (ΔmTSS) ≤0.5 units from baseline to Month 12
Total cost of RA-related treatment, in US dollars, at Month 6 | Baseline to 6 months
Total cost of RA-related treatment, in US dollars, at Month 12 | Baseline to 12 months

OTHER OUTCOMES:
Percentage of subjects with low disease activity (DAS28 <3.2) at Month 6 | Baseline to 6 months
Percentage of subjects with low disease activity (DAS28 <3.2) at Month 12 | Baseline to 12 months
Percentage of subjects with EULAR response at Month 6 | Baseline to 6 months
Percentage of subjects with EULAR response at Month 12 | Baseline to 12 months
Percentage of subjects with ACR50 response at Month 6 | Baseline to 6 months
Percentage of subjects with ACR50 response at Month 12 | Baseline to 12 months
Change in mTSS at Month 12 | Baseline to 12 months
Change in HAQ-DI score at Month 12 | Baseline to 12 months
Percentage of subjects with SAE | Baseline to 12 months
Change in work productivity as measured by the WPS-RA at Month 6 | Baseline to 6 months
Change in work productivity as measured by the WPS-RA at Month 12 | Baseline to 12 months
Change in health related QOL as measured by SF-36 at Month 6 | Baseline to 6 months
Change in health related QOL as measured by SF-36 at Month 12 | Baseline to 12 months
Change in health related QOL as measured by EQ-5D-5L at Month 6 | Baseline to 6 months
Change in health related QOL as measured by EQ-5D-5L at Month 12 | Baseline to 12 months
Percentage of subjects Incremental cost-effectiveness ratio (ICER) in terms of cost per QALY gained at Month 12 | Baseline to 12 months

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - Rheumatology Associates of North Alabama PC, Huntsville, Alabama
  - Dana Copeland Redyy Rheumatology, Chula Vista, California
  - Medvin Clinical Research, Covina, California
  - Western Connecticut Health Network, Danbury, Connecticut
  - Delaware Arthritis, Lewes, Delaware
  - Howard University, Washington D.C., District of Columbia
  - Robert W. Levin, MD, Clearwater, Florida
  - Arthritis Research Associates of Florida, Palm Harbor, Florida
  - Kenneth Stark, MD, Tavares, Florida
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Rheumatology Associates of Baltimore, Baltimore, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - June DO, PC, Lansing, Michigan
  - Beals institute PC, Lansing, Michigan
  - Shores Rheumatology, P.C., Saint Clair Shores, Michigan
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Timothy Kelly, MD, Las Vegas, Nevada
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Prospect Medical Offices Valley Medical Group, Midland Park, New Jersey
  - Overlook Medical Center Wound Healing Center, Summit, New Jersey
  - Rheumatology Associates of Long Island, Smithtown, New York
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Carolina Specialty Care, Statesville, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Paramount Medical Research, LLC, Middleburg Heights, Ohio
  - Southern Ohio Rheumatology, Wheelersburg, Ohio
  - Dr. Alan Kivitz, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - Carolina Health Specialist, Myrtle Beach, South Carolina
  - University of Tennesee Health Science, Memphis, Tennessee
  - Southwest Rheumatology Research LLC, Mesquite, Texas
  - Accurate Clinical Research, Nassau Bay, Texas
  - Arthritis Clinic of Central Texas, San Marcos, Texas
  - Arthritis Clinic of Northern VA, PC, Arlington, Virginia
  - Arthritis & Rheumatic Disease, Burke, Virginia
  - Western Washington Arthritis Clinic, Bothell, Washington
  - The Polyclinic, Seattle, Washington
  - Arthritis Northwest, P.L.L.C, Spokane, Washington
  - Gundersen Clinic, Ltd., Onalaska, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes